CLINICAL TRIAL: NCT06946303
Title: Identifying Key Attributes and Learning From a Local Falls Prevention Ambassador Programme
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Katie Robinson, Principal Research Fellow, University of Nottingham
Other Study IDs: FMHS-159-0324
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-04

CONDITIONS: Long Term Care
Keywords: long term care; falls
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic; Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Falls ambassador care home staff: Falls ambassador care home staff
  Interventions: Other: Survey; Other: Interview; Other: Observation

INTERVENTIONS:
Other: Survey — Pre and post survey on confidence and knowledge of falls
Other: Interview — Interview on the learning from the falls ambassador programme
Other: Observation — Observation of falls ambassador workshops

SUMMARY:
Managing falls for care home residents can be challenging for care home staff who work in complex settings and with residents with complex needs. Our previous research has identified that care homes would like more ongoing support and learning to improve their confidence in managing falls. One such programme is being set up in Lincolnshire.

The Lincolnshire Care Association are setting up a falls ambassador programme designed to provide ongoing support and learning for care homes on falls management. Exploring what this programme involves, what topics are covered and identified by care homes and whether they feel more confident in managing falls will help other areas in setting up similar programmes.

This research will explore the key attributes of the Lincolnshire Falls ambassador programme and explore whether it supports care home staff to feel more confident in managing falls by asking staff about their confidence before and after, observing the topics that are covered in the group meetings and by interviewing members of the programme after it has been established.

DETAILED DESCRIPTION:
To explore the key attributes of the Lincolnshire Falls ambassador programme and explore whether it supports care home staff to feel more confident in managing fall.

The following objectives will be achieved:

Describe the key activities of the programme. Identify the key themes of the discussions and shared learning. Explore whether care staff feel more confident in falls management. Identify barriers and facilitators to delivering the programme.

Survey: Pre and post survey of care home staff confidence. The survey will be distributed electronically using MS Forms by the programme leader at the start of the programme and after the programme. The survey will take up to 15 minutes to complete.

Interviews: Interviews with care home staff that have attended the programme to explore their learning and confidence. These will be undertaken face-to-face at a location convenient to the participant or over the telephone. With consent the interviews will be audio recorded and transcribed. If the participant prefers written field notes will be taken. The written transcripts and field notes will be classed as source data and retained. Any audit recording will be deleted to avoid retaining any personal identifiable information.

Observations: Observation of group meetings as part of the programme to identify the key areas of learning. The researcher will attend the meeting which will be either face-to-face or online. Field notes will be taken by the researcher and retained as source data.

ELIGIBILITY:
Inclusion Criteria:

* Any care home staff member attending the local falls ambassador programme

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Care home staff member attending the local falls ambassador programme
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Thematic analysis of learning from the programme | From enrolment to end of the falls ambassadors programme at 12 months
  Thematic analysis of learning from the programme

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Small number of participants